CLINICAL TRIAL: NCT05244629
Title: Copenhagen Mesenteric Stent Study - A Randomized Trial of Stent Versus Covered Stent Treatment for Chronic Mesenteric Ischemia
Acronym: COMESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Timothy Resch, Professor of Vascular Surgery, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 88754
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Mesenteric Ischemia; Bowel; Ischemic; Superior Mesenteric Atherosclerosis; Mesenteric Artery Stenosis; Stent Restenosis; Stent Occlusion; Stent Thrombosis; Stent-Graft Stenosis; Stent-Graft Thrombosis; Stent-Graft Restenosis
MeSH Terms: conditions — Mesenteric Ischemia; Ischemia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bare Metal Stent (Active Comparator)
  Interventions: Device: BMS vs. CS
- Covered Stent (Active Comparator)
  Interventions: Device: BMS vs. CS

INTERVENTIONS:
Device: BMS vs. CS — Patients will be randomized to treatment with either BeSmooth (BMS, Bentley Innomed GmBh) or BeGraft (CS, Bentley Innomed Gmbh)

SUMMARY:
Chronic mesenteric ischemia (CMI) is often caused by narrowings in the arteries providing blood to the intestines. Endovascular stent placement is considered the preferred treatment for this condition. Guidelines increasingly support the use of so called covered stents (CS) in stead of bare stents (BMS) for this use but the level of evidence for this is limited. Using CS incur additional costs for healthcare short-term but may prevent recurrence of narrowing and symptoms postoperatively benefitting patients and healthcare.

Study Objective:

To evaluate the outcomes after stenting of mesenteric arteries using BMS or CS.

Study Outcome:

Primary stent patency 1 year after placement

The trial will also evaluate complications, how often stents need to be reoperated, Quality of Life (QoL) and reasons for subjects death

Method:

This is a so called prospective, randomized controlled trial comparing CS vs. BMS. This means that one patients have agrred to treatment they will be randomly selected for treatment with either CS or BMS . The stent metal structure is identical in the two implants and the only difference is the graft covering, making this study unique.

The study will also collect blood samples for a biobank that will be used to study markers of disease and how these effect treatment outcomes.

All patients referred to the Department of Vascular Surgery due to CMI are considered for inclusion if they havechronic symptoms consistent with CMI, significant stenosis or occlusion of the superior mesenteric artery and are > 18 years Subjects not able to provide informed consent or who have non atherosclerotic cause of CMI, signs of acute loss of blood flow to the intestines cannot participate. Previous stent treatment in the superior mesenteric artery, pregnancy, allergies to contrast or stent materials are also reasons for not being included in this trial.

Side effects, risks and disadvantages for participants The risk for procedure-related complications is less than 5% and similar in both study groups. Most short-term complications are related to vascular access sites and consist of local bleeding and thrombosis. Other potential complications include impaired renal function due to contrast use, contrast allergy, arterial dissection and death.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic CMI of atherosclerotic or atherothrombotic etiology
* Intended endovascular treatment
* Symptoms consistent with CMI (pain, weight loss, diarrhea)
* Significant ostial stenosis (>50%) of the superior mesenteric artery on CTA
* Significant stenosis on angiography (>50% or >15mmHg pressure gradient)
* Patients > 18 years

Exclusion Criteria:

* No informed consent
* Non atherosclerotic cause of MI
* Acute mesenteric ischemia (AMI)
* Signs of acute bowel ischemia, peritonitis, laparotomy, sepsis
* Previous stent treatment in the superior mesenteric artery(ies)
* Target artery lesions >4cm in length
* Unable to cross lesion with guidewire
* Non-significant stenosis angiographically
* Pregnancy
* Allergies to contrast media or stent materials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients with open stents after 12 months | 12 months
  No evidence of occlusion, thrombosis or in-stent restenosis more than 30 percent

SECONDARY OUTCOMES:
Survival | 5 years
  reintervention free and overall survival
Quality of life accoring to SF 36 variables | 5 years
  SF 36

CONTACTS AND LOCATIONS:
Overall Officials: Timothy A Resch, MD, PhD, Principal Investigator — Deptarment of Vascular Surgery, Rigshospitalet
Locations (1):
- Department of Vascular Surgery, Heart Center, Copenhagen University Hospital - Rigshospitalet, København Ø, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brandtzag AA, Eiberg JP, Lonn L, Taudorf M, Resch TA. Copenhagen Mesenteric stent study (COMESS)-a randomized trial of stent versus covered stent treatment for chronic mesenteric ischemia. Trials. 2024 Jun 28;25(1):426. doi: 10.1186/s13063-024-08285-5. PMID 38943169